CLINICAL TRIAL: NCT06382051
Title: A Multicenter, Prospective, Study to Evaluate the Impact of Modifying the Validated Psoriasis Epidemiology Screening Tool (PEST) on the Potential Diagnosis of Psoriatic Arthritis in Adult Patients With Moderate-to-severe Plaque Psoriasis in Canada ("ScreenX")
Brief Title: Modifying PEST for Psoriatic Arthritis Screening
Acronym: ScreenX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CAIN457ACA06
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Plaque Psoriasis; Psoriatic Arthritis
Keywords: Psoriasis; Psoriatic Arthritis; PsA; Plaque Psoriasis; PsO; Implementation Science; Psoriasis Epidemiology Screening Tool
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEST Screening group (Other): When visiting their dermatologists, all eligible patients with moderate-to-severe plaque psoriasis (PsO) eligible for treatment with biologic Disease-Modifying Antirheumatic Drugs (bDMARDs) will be screened for psoriatic arthritis (PsA) using PEST+pictures+2, a variation of the PEST screening tool.
  The PEST+pictures+2 is made up of 3 components:
  1. Psoriasis Epidemiology Screening Tool (PEST) consisting of 5 simple questions
  2. PEST+2 refers to the PEST modified with two additional questions (Do you have morning stiffness that lasts for more than one (1) hour? Do you wake up at night because of low back or buttock pain?), AND
  3. PEST+pictures which provides an opportunity for patients to modify their answers to PEST questions 1, 3, and 5 by presenting them with pictures of swollen joints, fingernail pitting, and swollen fingers and toes.
  Interventions: Diagnostic Test: PEST Screening group

INTERVENTIONS:
Diagnostic Test: PEST Screening group — PEST Screening group

SUMMARY:
The purpose of this study is to assess the impact of adding two questions and pictures to the validated PEST on the potential diagnosis of PsA in participants with moderate-to-severe plaque PsO in Canada.

DETAILED DESCRIPTION:
Patients will be enrolled in the study for up to 66 days and will be asked to fill-out a PsA screening questionnaire at their first dermatologist visit. Patients screening positive for PsA will have a second visit with a rheumatologist where a full PsA diagnosis assessment will be performed. A remote 'end of study' (EOS) visit will be conducted by the dermatologist to document the patient's biologic Disease-Modifying Antirheumatic Drugs (bDMARDs) treatment choice and status.

ELIGIBILITY:
Key inclusion criteria:

1. Moderate-to-severe plaque PsO patients who are candidates for bDMARDs, as per provincial reimbursement criteria
2. Adult patients at the time of informed consent signature
3. Patients able to understand and willing to comply with protocol requirements, instructions, and restrictions
4. Residents of Canada

Key exclusion criteria:

1. Patients who have previously screened positive for PsA through PEST or any other screening method
2. Patients who have been diagnosed with PsA and/or followed by a rheumatologist
3. Patients who have been diagnosed with inflammatory arthritis unrelated to PsA (rheumatoid arthritis, reactive arthritis, enteropathic arthritis, axial spondyloarthritis)
4. Patients treated with a bDMARD for moderate-to-severe plaque PsO or any other medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) for PEST and PEST+2 in adult patients with moderate-to-severe plaque PsO who are candidates for bDMARDs | Up to approximately 1 year
  To assess the impact of adding two questions (morning stiffness and low back or buttock pain) to the validated PEST for the potential diagnosis of PsA in moderate-to-severe plaque PsO patients who are candidates for biologic disease-modifying antirheumatic drugs (bDMARDs) The primary clinical question of interest is: Can the addition of two questions to PEST pertaining to presence of morning stiffness and low back or buttock pain (i.e., PEST+2) allow for improved screening and diagnosis of PsA in patients with moderate-to-severe plaque PsO?

SECONDARY OUTCOMES:
Proportion of patients scoring negative on PEST and positive on PEST+2 with a confirmed new PsA diagnosis or suspicion of PsA by a rheumatologist | Up to approximately 1 year
  To estimate the proportion of patients with a confirmed or suspected PsA diagnosis referred by dermatologists using PEST+2 only
Proportion of patients with a confirmed new PsA diagnosis or suspicion of PsA by a rheumatologist | Up to approximately 1 year
  Proportion of patients with a new PsA diagnosis or suspicion of PsA, confirmed by the rheumatologist who scored:
  1. Negative on PEST and positive on PEST+pictures
  2. Negative on PEST+2 and positive on PEST+pictures+2 will be evaluated to assess the impact of adding pictures as reference to guide patients answering the screening questions (question 1, 3, and 5)
Proportion of patients with a false positive score between each group | Up to approximately 1 year
  Proportion of patients with false positive score between each group will be evaluated:
  1. PEST+2 vs. PEST+pictures+2
  2. PEST+pictures vs. PEST
  3. PEST+pictures+2 vs. PEST
Description of the baseline characteristics of the positive screening score and negative screening score patients for both PEST and PEST+2 tests | Up to approximately 1 year
  Description of the baseline characteristics (i.e., patient age, biological sex, years since plaque PsO diagnosis, medical history, disease characteristics, concomitant treatments, height, weight, etc.) of the positive screening score and negative screening score patients for both PEST and PEST+2 tests will be evaluated to determine patient's baseline characteristics.
Patient acceptability/user experience of the PEST+2 questionnaire | Up to approximately 1 year
  Summary scores of the patient acceptability questionnaire of PsA screening questionnaires and a categorical presentation of question-by-question responses at Visit 1
Administration of dermatologist quantitative surveys | Up to approximately 1 year
  Administration of dermatologist quantitative surveys, as well as open-ended qualitative questions to assess the acceptability and feasibility of the PEST+pictures+2 from the perspective of dermatologists
Qualitative interview with selected dermatologists | Up to approximately 1 year
  Brief 1:1 qualitative interview with selected dermatologists (maximum 12) to assess their knowledge, beliefs, and attitudes towards PsA screening (e.g., motivation to screen)
Intervention Appropriateness Measure (IAM) | Up to approximately 1 year
  To assess the appropriateness of the PEST+2 from the perspective of rheumatologists

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Canada (10):
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Fredericton, New Brunswick
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Richmond Hill, Ontario
  - Novartis Investigative Site, Stoney Creek, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.